CLINICAL TRIAL: NCT02747381
Title: The Effect of Vitamin D Supplementation on the Pulmonary Functions of Adult Asthmatic Egyptian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amani Mohamed, Teaching assisstant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (1122)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — alfacalcidol; Hydroxycholecalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): receive Alfacalcidol 1 mcg daily for 4 months beside the conventional asthma medications
  Interventions: Dietary Supplement: Alfacalcidol
- control (No Intervention): Asthmatic patients receiving conventional asthma medications

INTERVENTIONS:
Dietary Supplement: Alfacalcidol — 1-alpha hydroxy cholecalciferol 1 mcg
  Other Names: One alpha
  Arms: intervention

SUMMARY:
This study evaluates the effect of vitamin D supplementation in the form of Alfacalcidol on the the pulmonary function of adult asthmatic Egyptian patients

DETAILED DESCRIPTION:
Asthmatic patients are recruited and divided into two groups. One receives Alfacalcidol beside their normal medications while the other acts as a control group receiving the normal asthma medication.

Both groups are followed up for four months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with asthma
2. Non-smokers

Exclusion Criteria:

1. Liver impairment
2. Kidney impairment
3. Patients receiving digoxin
4. Known hypersensitivity to 1α-hydroxyvitamin D3, vitamin D or any of its analogues and derivatives
5. Hypercalcaemia
6. Hyperphosphatemia
7. Pregnancy and breast-feeding
8. Patients on nutritional supplements with a potential effect on 25(OH)D serum concentrations
9. Had a History of stones in the urinary tract or diseases of calcium or bone metabolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
forced expiratory volume % predicted values | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Amani Ali, Principal Investigator — Faculty of pharmacy, Cairo university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ali AM, Selim S, Abbassi MM, Sabry NA. Effect of alfacalcidol on the pulmonary function of adult asthmatic patients: A randomized trial. Ann Allergy Asthma Immunol. 2017 May;118(5):557-563. doi: 10.1016/j.anai.2017.02.014. Epub 2017 Apr 1. PMID 28377173